CLINICAL TRIAL: NCT07067190
Title: Clinical and Radiographic Evaluation of Mandibular Implant Assisted Overdenture Between Bar Attachment and Bar With OT Cap Attachment: Randomized Control Clinical Trial
Brief Title: Mandibular Implant Overdenture With OT Cap Bar vs Bar Attachment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maisa Mohamed Farid Shaaban (Other)
Responsible Party: Sponsor-Investigator, Maisa Mohamed Farid Shaaban, PhD Candidate, Department of Prosthodontics, Faculty of Oral and Dental Medicine, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MF-OTBarRCT2024
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Edentulous Mandible; Implant-Supported Overdentures
Keywords: Bar Attachment; OT Cap Attachment; Implant-Assisted Overdenture; Dental Implants; Mandibular Denture Retention; Crestal Bone Loss; Patient Satisfaction; Attachment Wear
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled clinical trial comparing bar-only attachment vs. bar with OT Cap attachment in mandibular implant-supported overdentures.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor (statistician) will be blinded to group allocation to reduce assessment bias. Neither the participant nor the care provider can be blinded due to the visible nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bar Attachment Group (Active Comparator): Participants in this group will receive mandibular implant-supported overdentures retained by a conventional cast bar attachment. Three implants will be placed in the anterior mandible (midline and canine positions), and a single bar will be fabricated and attached to the implants. The overdenture will be adjusted to fit over the bar with no additional retentive components. This group represents the standard treatment modality for implant-retained overdentures.
  Interventions: Device: Conventional Bar Attachment
- Bar with OT Cap Attachment Group (Experimental): Participants in this group will receive mandibular implant-supported overdentures using a bar combined with two OT Cap (sphere) attachments for added retention. The same implant placement protocol will be followed as in the comparator group. The bar will include OT Cap housings, and the overdenture will be relined to incorporate the corresponding female caps. This intervention is designed to improve denture retention, reduce component wear, and enhance patient satisfaction.
  Interventions: Device: Bar with OT Cap Attachment

INTERVENTIONS:
Device: Conventional Bar Attachment — A rigid cast bar attachment fabricated and screwed onto three mandibular implants (placed at the midline and canine areas). The bar connects the implants to provide splinting and retention for a mandibular overdenture without the use of additional retentive components such as OT Caps. The overdenture is adjusted to fit passively over the bar and picked up intraorally.
  Arms: Bar Attachment Group
Device: Bar with OT Cap Attachment — A cast bar attachment fitted with two OT Cap attachments, which are designed to improve prosthesis retention and load distribution. This bar system is installed on three mandibular implants (midline and canine regions). The mandibular overdenture is relined to incorporate the female retentive caps that snap onto the OT Caps. This system combines the splinting benefits of the bar with the resilient retention of stud attachments.
  Arms: Bar with OT Cap Attachment Group

SUMMARY:
This clinical study is being conducted at Cairo University to evaluate two different types of attachments used with implant-supported dentures in the mandible. Patients who have lost all their teeth in the lower jaw receive implants to help hold their dentures in place. This study compares two types of attachments for connecting the denture to the implants:

1. Bar attachment only, which is a traditional method.
2. Bar with OT Cap attachment, which is a newer design that includes a small sphere (cap) to help with retention and comfort.

The purpose of this study is to find out which attachment type works better in terms of:

1. How well the denture stays in place (retention)
2. How much bone is lost around the implants over time (crestal bone loss)
3. How much the attachment parts wear out (cap wear)
4. How satisfied the patients are with their dentures

The study is a randomized controlled trial. This means participants will be randomly assigned to one of the two groups (bar-only or bar with OT Cap). All participants will receive complete dentures and three dental implants in the lower jaw.

Follow-up will include measurements of denture retention and cap wear at the time the denture is inserted and again after 6 months. Bone loss will be checked with digital X-rays, and patient satisfaction will be assessed using a short questionnaire.

The study will include 22 participants (11 in each group), aged 30 to 65, who are healthy and have enough bone in the jaw to support implants.

This study is designed to help dentists and patients make better decisions about which type of implant attachment provides better long-term results and patient comfort.

DETAILED DESCRIPTION:
This randomized controlled clinical trial is designed to evaluate and compare the clinical and radiographic outcomes of two mandibular implant-supported overdenture attachment systems: (1) conventional bar attachment, and (2) bar with OT Cap (sphere) attachment. The objective is to determine which system provides superior performance in terms of prosthesis retention, crestal bone preservation, attachment wear, and patient satisfaction.

A total of 22 completely edentulous participants, aged between 30 and 65 years and meeting strict inclusion criteria, will be enrolled. Each participant will receive three endosseous implants placed in the anterior mandibular region (midline and canine positions). Following a four-month osseointegration period, participants will be randomly allocated (1:1) to one of two intervention groups: Group A (bar attachment only) and Group B (bar with OT Cap sphere attachments).

The prosthetic protocol involves the fabrication and delivery of maxillary and mandibular complete dentures, followed by intraoral placement and pick-up of the attachment systems. The primary outcome is denture retention, assessed at baseline (T0) and after 6 months (T6) using a digital force gauge. Secondary outcomes include crestal bone loss (evaluated via standardized digital radiographs), cap wear (measured using electron microscopy), and patient satisfaction (assessed using a validated Visual Analog Scale questionnaire).

Randomization will be conducted using a computer-generated sequence with allocation concealment ensured via opaque sealed envelopes. Due to the nature of the intervention, blinding of participants and clinicians is not feasible; however, outcome assessment and statistical analysis will be performed by a blinded examiner.

This study addresses a critical gap in the comparative assessment of attachment systems for implant-retained mandibular overdentures. While bar attachments are widely used for their rigidity and implant splinting capacity, recent innovations such as the OT Cap aim to enhance retention and reduce maintenance through added resilience. By directly comparing these two configurations in a controlled setting, the study aims to contribute clinically relevant data to guide prosthodontic treatment planning for edentulous patients.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous healthy patients
* Age between 30 and 65 years
* Adequate bone volume in the anterior and premolar-molar region (minimum 11 mm)
* Adequate inter-arch space (12-14 mm)

Exclusion Criteria:

* Severe maxillomandibular skeletal discrepancy
* Parafunctional habits (e.g., clenching, bruxism)
* Temporomandibular joint disorders
* Heavy smokers (≥20 cigarettes/day)
* History of head and neck radiation
* History of chemotherapy
* Systemic conditions that may interfere with healing or bone quality (e.g., uncontrolled diabetes, osteoporosis, bisphosphonate therapy)
* Drug abuse or alcohol dependence

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Retention of Mandibular Implant-Supported Overdenture | Baseline (T0) and 6 months after overdenture insertion (T6)
  Retention will be measured using a digital force gauge that applies a vertical dislodging force to the mandibular overdenture. The force required to dislodge the denture from the attachments will be recorded in Newtons. Measurements will be performed at two time points: at the time of prosthesis insertion (T0) and six months post-insertion (T6). The retention values will be used to compare the effectiveness of bar-only versus bar with OT Cap attachment systems.

SECONDARY OUTCOMES:
Crestal Bone Loss Around Implants | Baseline (T0) and 6 months after overdenture insertion (T6)
  Crestal bone levels will be assessed using standardized digital radiographs with the Digora long-cone parallel technique. Measurements will be taken from the implant shoulder to the first bone-to-implant contact point on mesial and distal surfaces. The difference in bone height between baseline (T0) and six months (T6) will be calculated in millimeters to determine bone loss.
Attachment Cap Wear | Baseline (T0) and 6 months after overdenture insertion (T6)
  Cap wear will be evaluated by measuring the internal diameter changes of the OT Cap components using scanning electron microscopy (SEM). Measurements will be taken at baseline (T0) and after 6 months (T6) to assess material degradation and fit deterioration.
Patient Satisfaction with Overdenture | 6 months after overdenture insertion (T6)
  Patient satisfaction will be assessed using a validated Visual Analog Scale (VAS) questionnaire that evaluates comfort, stability, appearance, chewing ability, speech, ease of cleaning, and overall satisfaction. Each parameter is rated from 0 (not satisfied at all) to 100 (completely satisfied). The results will be used to compare the perceived outcomes between the two intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Maisa MF Shaaban Gomaa, PhD candidate, Principal Investigator — Faculty of Oral and Dental Medicine, Cairo University; Hamdy Abo El-Fotouh, Professor, Study Chair — Faculty of Oral and Dental Medicine, Cairo University; Noha Ali, Assistant Professor, Study Director — Faculty of Oral and Dental Medicine, Cairo University; Ahmed Hamed, Lecturer, Study Director — Faculty of Oral and Dental Medicine, Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study is self-funded and conducted as part of a doctoral thesis project. No data-sharing mechanism or repository has been established, and participants were not consented for external data sharing. Additionally, confidentiality and ethical guidelines limit redistribution of participant-level data